CLINICAL TRIAL: NCT06216613
Title: Testing Effects of Swim Instruction on Autistic Children's Swimming and Water Safety Skills
Brief Title: Testing Swim Instruction for Autistic Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: FP00000742
Record Dates: First submitted 2024-01-11; First posted 2024-01-22 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Autism
Keywords: Autism; Water Safety; Swimming
MeSH Terms: conditions — Autistic Disorder

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial with 50 participants who will be randomized 1:1 to either the Sensory Enhanced Aquatics intervention or control condition with standard swim lessons.
Who Masked: Outcomes Assessor
Masking Description: The nature of our intervention precludes blinding of the interventionists and participants; however, investigators not involved in the intervention, data analysts and research assistants will be blinded to condition.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sensory Enhanced Aquatics (Experimental): Sensory Enhanced Aquatics is a specialized swimming and water safety program for autistic children.
  Interventions: Behavioral: Sensory Enhanced Aquatics
- Standard Swim Lessons (Active Comparator): Standard swim lessons which are provided to the general public will be used as the comparison group.
  Interventions: Behavioral: Standard Swim Lessons

INTERVENTIONS:
Behavioral: Sensory Enhanced Aquatics — Sensory Enhanced Aquatics (SEA) utilizes the Sensory Profile to individualize lessons based on children's sensory preferences. The program incorporates evidence-based approaches for autistic children, including: 1) visual supports, 2) sensory supports, 3) communication strategies, 4) behavioral strategies, and 5) modeling to maximize skill acquisition. Lessons will be 1:1 with social opportunities at the beginning and end of each lesson. Like standard swim lessons, skills are taught in progression from water orientation (e.g., blowing bubbles, submerging different body parts) to advanced swimming (e.g., swimming 15 or more yards of different swim strokes). All lessons include instruction of water safety skills. Each skill has been task analyzed by therapists so instruction can be graded according to children's ability. A social story is provided to transition children to lessons. SEA curriculum was reviewed by USA Swimming Foundation and is included as a Swim Lesson Network Provider.
  Arms: Sensory Enhanced Aquatics
Behavioral: Standard Swim Lessons — Standard swim lessons will adhere to USA Swimming Foundation Swim Network Provider requirements ensuring lessons meet or exceed industry best practices. Lessons have up to a 1:5 instructor to child ratio and will focus on stroke development and water-safety with skills advancing from water-orientation to stroke technique and endurance.
  Arms: Standard Swim Lessons

SUMMARY:
The goal of this clinical trial is to compare the effects of a specialized swimming and water-safety program (Sensory Enhanced Aquatics) and standard swimming lessons for autistic children. The main question[s]it aims to answer are:

* Do Sensory Enhanced Aquatics and standard swimming lessons improve swimming and water-safety skills of autistic children?
* Which participant characteristics are associated with the highest post-intervention swim skills and water safety across both groups?

Participants will:

* Complete questionnaires, motor, and swim tests before the intervention.
* participate in 16, 30-minute Sensory Enhanced Aquatics lessons.
* Complete a swim test after the intervention.
* Complete an interview. Researchers will compare with participation in standard swim lessons to see if which bests teaches swimming and water-safety to autistic children.

DETAILED DESCRIPTION:
The investigators will conduct a single blind, randomized controlled pilot trial to test the differential effects of an eight-week (16 lesson) Sensory Enhanced Aquatics intervention and standard swim lessons on attainment of swimming and water safety skills of autistic children. Investigators will enroll 50 autistic children aged 5-9 years who will be randomized 1:1 by minimization to either the Sensory Enhanced Aquatics intervention or standard swim lessons to minimize imbalanced group allocation by autism severity and baseline swim skill. Aim 1 will compare the effects of Sensory Enhanced Aquatics to standard swimming lessons on swimming and water safety skills of autistic children with a swim test based on Red Cross water competency guidelines. Aim 2 will assess which participant characteristics (e.g., age, motor ability, autism severity) are associated with the highest post-intervention swim skills and water safety across both groups to inform who benefits most from swim instruction. Child sex and co-occurring motor impairment will be considered as potential covariates. Data will be collected before swim lessons and after 8 weeks of Sensory Enhanced Aquatics or standard lessons. The investigators hypothesize children in both groups will demonstrate improvement in swimming and water safety skills with greater improvements in the Sensory Enhanced Aquatics group; autism severity and motor ability will have the greatest associations with swim skill in both groups. Our exploratory aim will employ post-intervention semi-structured interviews to explore child, parent, and instructor perspectives about instructional methods most effective for developing swimming and water-safety among autistic children. The information obtained from this study will improve our understanding of the best strategies for swim instruction for autistic children and support our long-term goal to make Sensory Enhanced Aquatics scalable on the national level to prevent drowning of autistic children.

ELIGIBILITY:
Inclusion Criteria:

* Age 5-9 yrs. who have received a clinical diagnosis for autism based on Diagnostic and statistical manual of mental disorders: DSM-5 criteria
* A Social Responsiveness Scale-2 (SRS-2) T-score of ≥ 60
* Sufficient functional ability to understand directions and communicate preferences (verbally or non-verbally)
* Baseline swim test score ≤22
* No plans to relocate outside the study area during the intervention period.
* Physician consent.

Exclusion Criteria:

* Uncontrolled epilepsy, as seizures increase risk of drowning.
* Baseline swim test score ≥23
* Aggressive behaviors that would put instructor safety at risk.

Ages: 5 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 51 (Actual)
Dates: Start 2024-04-14 (Actual); Primary Completion 2025-07-30 (Actual); Study Completion 2025-09-04 (Actual)

PRIMARY OUTCOMES:
Child Swim Test | pre and post 8 weeks
  Individual performance test of 5 American Red Cross water competency skills, 5 preparatory swim skills and 2 water-safety skills scored on a 4-point scale with total scored ranging from 0-38.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: Yes
The raw data will be preserved at the local site per local institutional policies and guidelines. However, the data that will be preserved and made available for sharing will be the summary or scored data for each participant at each data collection timepoint. We have made this decision to provide summary or scored data to allow for the data that are available to be consistent across the various uses (e.g., to minimize the likelihood of scoring errors by others who may use the data). However, if the study sponsor or other regulatory entity requests that we reconsider this decision, we are willing to consider this request. We will also share audio recordings of interviews.
Supporting Information: Study Protocol, ICF, Analytic Code
Time Frame: The data will be made available no later than the time of an associated publication or at the end of the performance period, whichever comes first. We will also work closely with our Data and Safety Monitoring Board to identify any applicable embargo periods that may be necessary to maintain the integrity of the study and will implement these in an appropriate manner that is consistent with NIH and local institutional policies. The data provided to the repository will be available indefinitely while that repository continues to exist.
Access Criteria: we will upload our data to the National Database for Autism Research (NDAR)
URL: https://www.nih.gov/health-information/nih-clinical-research-trials-you/personal-stories/researcher-story-national-database-autism-research-ndar